CLINICAL TRIAL: NCT00379990
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Investigate the Safety, Tolerability, Pharmacokinetics and Effect on Synovial Thickness and Vascularity of 28 Days Repeat Dosing of GW274150 or 7.5mg Prednisolone in RA Subjects.
Brief Title: A Study To Investigate GW274150 Or Prednisolone In Rheumatoid Arthritis Taken Repeatedly For 28 Days.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RA4104917
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Arthritis, Rheumatoid
Keywords: iNOS; Exhaled NO; Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GW 274150; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- GW274150 60 mg once daily for 28 days (Experimental): 60 mg GW274150 taken once daily for 28 days
  Interventions: Drug: GW274150
- Prednisolone 7.5 mg once daily for 28 days (Active Comparator): 7.5 mg prednisolone taken once daily for 28 days
  Interventions: Drug: Prednisolone
- Placebo once daily for 28 days (Placebo Comparator): Placebo taken once daily for 28 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GW274150 — 60 mg /day
  Arms: GW274150 60 mg once daily for 28 days
Drug: Prednisolone — 7.5 mg/day
  Arms: Prednisolone 7.5 mg once daily for 28 days
Other: Placebo — Placebo
  Arms: Placebo once daily for 28 days

SUMMARY:
This is an exploratory study to examine the effect of iNOS inhibition in rheumatoid arthritis patients. The study involves 28 days repeat dosing with GW274150 (dose determined by the results from a previous study), prednisolone (7.5mg) or placebo.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of rheumatoid arthritis according to the revised 1987 criteria of the American College of Rheumatology
* Female subjects who are not capable of becoming pregnant
* Active disease defined as Disease Activity Score (DAS) 28 = 4.0 and at least one metacarpal-phalangeal finger (MCP) joint with either detectable vascularity or thickness
* Stable doses of disease modifying anti-rheumatic drugs (DMARDs), (which can include but is not restricted to methotrexate, sulphasalazine and hydroxychloroquine in any combination) for 8 weeks prior to enrollment
* Patients receiving methotrexate must be on stable folate supplements
* Must have been on stable doses for 2 weeks prior to screening if using COX inhibitors
* Signed consent form
* The patient is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions

Exclusion criteria:

* The subject is using, or has used, oral glucocorticoids within 8 weeks of enrollment
* The subject is currently receiving anti-rheumatic biological therapy (e.g. infliximab, adalimumab, etanercept or anakinra)
* The subject received their final dose of infliximab or adalimumab within 3 months of enrollment
* The subject received their final dose of etanercept or anakinra within 1 month of enrollment
* The subject has received another investigational drug within 30 days
* The subject drinks more than 28 units (male) or 21 units (female) of alcohol in a week
* History of liver or renal disease in the 6 months prior to screening
* The subject has a history of drug or other allergy
* Subject is positive for Hepatitis B and C or HIV virus
* The subject has positive pregnancy test
* The subject has positive test for drugs of abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Measurment of synovial vascularity | Day 1, Day 15 and Day 28
  Power Doppler ultrasonographic measurement of synovial vascularity

SECONDARY OUTCOMES:
Synovial thickness | Day 1, 15 and 28
  High frequency ultrasound measurement of synovial thickness
Safety: ECG | Day 1, 15 and 28
  12-lead ECG meaurements
Safety: Vital Signs | Day 1, 15 and 28
  Blood pressure and heart rate
Safety: Laboratory | Day 1, 8, 15, 22, 28 and Follow Up
  Laboratory assessments including liver function tests, amylase and lipase
Pharmacokinetics: Cmax | Day 15 and Day 28
  Maximum plasma concentration of GW274150
Pharmacokinetics: Trough | Days 8,15 and Day 28
  Trough plasma concentration of GW274150
Tolerability | Day 1 to Day 28 and Follow Up
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Belgrade, Serbia
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Seymour M, Petavy F, Chiesa F, Perry H, Lukey PT, Binks M, Donatien PD, Freidin AJ, Eckersley RJ, McClinton C, Heath K, Prodanovic S, Radunovic G, Pilipovic N, Damjanov N, Taylor PC. Ultrasonographic measures of synovitis in an early phase clinical trial: a double-blind, randomised, placebo and comparator controlled phase IIa trial of GW274150 (a selective inducible nitric oxide synthase inhibitor) in rheumatoid arthritis. Clin Exp Rheumatol. 2012 Mar-Apr;30(2):254-61. Epub 2012 Apr 13. PMID 22409880